CLINICAL TRIAL: NCT00052013
Title: A Phase II Open-Label Study of Oral, Continuous, Once Daily PTK787/ZK 222584 in Patients With Von Hippel-Lindau Disease (VHL) and Hemangioblastoma (HB)
Brief Title: Treatment of Von Hippel-Lindau (VHL)-Related Hemangioblastoma With PTK787/ZK 222584
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPTK787 0144
Record Dates: First submitted 2003-01-21; First posted 2003-01-22 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2011-02

CONDITIONS: Von Hippel-Lindau Disease; CNS Hemangioblastoma; Retinal Hemangioblastoma
Keywords: von Hippel-Lindau disease,; CNS,; hemangioblastoma,; retinal
MeSH Terms: conditions — von Hippel-Lindau Disease; Hemangioblastoma | interventions — vatalanib

ARMS (1):
- PTK787/ZK 222584 (Experimental)
  Interventions: Drug: PTK787/ZK 222584

INTERVENTIONS:
Drug: PTK787/ZK 222584

SUMMARY:
The purpose of this study is to determine whether PTK787/ZK 222584 is effective in treating hemangioblastoma of the brain and/or retina in patients with von Hippel-Lindau disease. The study will also assess safety and tolerability of PTK787/ZK 222584, and changes in markers of angiogenesis (new blood vessel growth).

ELIGIBILITY:
Inclusion criteria:

* Confirmed diagnosis of VHL disease
* One or more measurable CNS hemangioblastoma, if symptomatic, must be refractory or not amenable to standard therapy, if asymptomatic, must have had at least one prior neurosurgical treatment/ procedure; and/or: at least one untreatable or treatment-refractory retinal hemangioblastoma that is causing impaired visual function
* Karnofsky Performance Status >=60
* Life expectancy > 3 months
* Able to sign informed consent
* Adequate hematologic status, liver and kidney function

Exclusion criteria:

* Patients with other VHL-related tumors requiring or amenable to standard treatment
* Severe or uncontrolled concurrent illnesses that could compromise participation in the study
* Total urinary protein in 24 hour collection > 500 mg
* Pregnant or breast feeding females, adults of reproductive potential not using effective contraception (hormonal methods not considered effective due to possible decreased effectiveness secondary to drug interaction with PTK787). Women of childbearing potential must have negative serum pregnancy test prior to initiation of treatment.
* Acute or chronic liver disease
* Diagnosis of HIV infection
* GI function that may alter absorption of PTK787
* Patients taking coumadin (warfarin sodium)
* Prior therapies (investigational drugs, chemotherapy) within 4 weeks prior to study entry
* Prior therapies (biologic, hormonal, immunotherapy, radiation therapy, surgery) within two weeks prior to study entry.
* Patients unwilling or unable to comply with protocol requirements
* Patients with concurrent, non VHL-related malignancies other than non-melanoma skin cancer
* Patients with contraindication to MRI imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2003-02; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Evaluate efficacy

SECONDARY OUTCOMES:
Evaluate changes in dynamic contrast enhanced magnetic resonance imaging
To explore the correlation of the pharmacokinetics
To assess changes in surrogate markers of angiogenesis

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina